CLINICAL TRIAL: NCT01545024
Title: Effect of DPP-IV Inhibitor on Glycemic Control and Autonomic Neuropathy in Adult Patients With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, Investigator, Nagaoka Red Cross Hospital
Other Study IDs: 4-Kamoi
Record Dates: First submitted 2012-02-23; First posted 2012-03-06 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DPP-IV inhibitor
  Interventions: Drug: Sitagliptin, 50 mg once per day per os

INTERVENTIONS:
Drug: Sitagliptin, 50 mg once per day per os — Before and one year after treatment with DPP-IV inhibitor in diabetic patients with AND.
  Other Names: Nothing

SUMMARY:
Rocca et al. reported first that the secretion of incretins, particular GLP-1 in rat is regulated by the enteric nervous system, the afferent and efferent vagus nerves [1]. Further, Kazakos et al. [2] reported that autonomic nerve disturbance (AND) in patients with T2DM impaired the incretin effect owing to decreased GLP-1 secretion. However, Toft-Nielsen et al. [3] reported that the decreased GLP-1 responses in the patients with type 2 diabetes mellitus (T2DM) are unlikely to be related to the AND and, thus, did not support the results of Rocca et al. and Kazakos et al. Recently, Yabe at al. [4] also observed the same observations in Japanese patients with T2DM. Meanwhile, Jin et al. reported that administration of DPP-IV inhibitor recovered the disturbance of diabetic nerve dysfunction in rat [5]. However, it is unknown whether the administration of DPP-IV inhibitor effects on the AND in human, although many studies are performed to investigate the effect of the DPP-IV inhibitors on glycemic control.

Accordingly, it is significant to reinvestigate an effect of DPP-IV inhibitor on glycemic control and autonomic neuropathy in diabetic patients.

DETAILED DESCRIPTION:
Autonomic nerve disturbance (AND) is estimated to use coefficient of variance of electrocardiographic beat-to-beat intervals (C.V. R-R). Maximal change of the C,V. R-R with from usual breathing to deep breathing at the resting was used for the evaluation of AND. Less than 2.0 % of the maximal value is estimated to have a positive to AND.

Glycemic control is estimated to measure change of HbA1c value once three months per year.

ELIGIBILITY:
Inclusion Criteria:

type 1 and 2 diabetes mellitus patients

* Patients who have AND determined by C.V. R-R.
* Outpatients regularly visiting hospital
* Patients 20 years old (gender is disregarded)

Exclusion Criteria:

Patients with a serious complication in the heart, liver or kidney

* Pregnant or possibly pregnant patients, or lactating patients
* Patients complicated with a malignant tumor at present.
* Patients participating in other clinical study.
* Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 and 2 diabetic patients who have AND determined by C.V. R-R, outpatients regularly visiting hospital and more than 20 years old (gender is disregarded). Type 1 diabetic patients are treated with Epalrestat 50 mg. 150 mg t.i.d., while type 2 diabetic patients are treated with DPP-IV inhibitors.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | For one year after treatment wih DPP-IV inhibitor
  As marker of HbA1c

SECONDARY OUTCOMES:
autonomic nerve disturbance | Before and one year after treatment with DPP-IV inhibitor
  Before and after measurment with R-R CV in ECG at rest and respiratory deeping

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital
Locations (1):
- Nagaoka Red Cross Hospital, Nagaoka, Niigata, Japan

REFERENCES:
- [Background] 1. Rocca AS, Brubaker PL. Role of the vagus nerve in mediating proximal nutrient-induced glucagon-like peptide-1 secretion. Endocrinology 1999;140:1687-1694. 2. Kazakos KA, Sarafidis PA, Yovos JG. The impact of diabetic autonomic neuropathy on the incretin effect. Med Sci Monit 2008; 14:CR213-220. 3. Toft-Nielsen MB, Damholt MB, Madsbad S, Hilsted LM, Hughes TE, Michelsen BK, Holst JJ. Determinants of the impaired secretion of glucagon-like peptide-1 in type 2 diabetic Patients. J Clin Endocrinol Metab 2001;86:3717-3723. 4. Yabe D, Watanabe K, Sugawara K, Kuwata H, Kitamoto Y, Sugizaki K, Fujiwara S, Hishizawa M, Hyo T, Kuwabara K, Yokota K, Iwasaki M, Kitatani N, Kurose T, Inagaki N, Seino Y (2011) Comparison of incretin immunoassays with or without plasma extraction: incretin secretion in Japanese patients with type 2 diabetes. J Diabetes Invest 2011;2:DOI. 5. Jin HY, Liu WJ, Park JH, Baek HS, Park TS. Effect of dipeptidyl peptidase-IV (DPP-IV) inhibitor (Vildagliptin) on peripheral nerves in streptozotocin-induced diabetic rats. Arch Med Res 2009;40:536-544.